CLINICAL TRIAL: NCT06218381
Title: The Effects of Very Brief Exposure on PTSD in U.S. Combat Veterans
Acronym: PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Bradley Peterson, Chief, Division of Child & Adolescent Psychiatry, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHLA-20-00782
Record Dates: First submitted 2024-01-09; First posted 2024-01-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder; Veteran; Very Brief Exposure
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Image Exposure Arm (Experimental): This within-subjects design study will have all participants view three types of exposure during fMRI scanning: VBE to combat images, VBE to masked everyday scenes (control), and conscious visible exposure to the same images (control).
  Interventions: Other: Very Brief Exposure to Combat Images

INTERVENTIONS:
Other: Very Brief Exposure to Combat Images — In VBE, a series of pictures representing a person's fears (e.g., a combat scene with arousing visuals) is presented very briefly (17 ms), followed by a masking stimulus that prevents conscious recognition of each picture. This sequence of picture-mask stimuli is repeated many times in an exposure session.

SUMMARY:
The goal of this clinical trial is to develop a new behavioral treatment for U.S. combat veterans with post-traumatic stress disorder (PTSD), very brief exposure to combat-related stimuli. The main questions it aims to answer are:

1. How does Very Brief Exposure (combat images and control everyday images) and Visible Exposure to combat stimuli affect brain activity and subjective fear ratings?
2. To what extent are participants aware of the stimuli presented and tolerating the exposures?

All participants will view both very brief exposure and visible exposure to combat stimuli in the functional magnetic brain imaging (fMRI) scan. They will provide ratings of fear, awareness, and tolerability. Researchers will compare U.S. combat veterans with PTSD and healthy controls to confirm differences in brain region activation and ratings.

DETAILED DESCRIPTION:
The prevailing treatment for Post-traumatic Stress Disorder (PTSD) is exposure: the confrontation of traumatic memories, in one form or another. Although exposure therapies are effective for combat related PTSD, confronting traumatic memories is inherently aversive, which may contribute to problems with patient acceptance. For example, trauma-focused PTSD therapies have higher dropout rates than non-trauma-focused therapies, and combat vets who drop out in real-world practice have more avoidance behaviors and greater arousal than those who remain in treatment. Study investigators have developed an alternative form of exposure that has been repeatedly shown to reduce behavioral, physiological, and self-reported fear symptoms in phobic persons without having them directly confront feared situations, and thus without causing them to experience emotional distress. In Very Brief Exposure (VBE), a series of pictures representing a person's fears (e.g., a combat scene with arousing visuals) is presented very briefly (17 ms), followed by a masking stimulus that prevents conscious recognition of each picture. This sequence of picture-mask stimuli is repeated many times in an exposure session.

The goal is to develop a new behavioral treatment for U.S. combat veterans with PTSD, VBE to combat-related stimuli by:

1. Identifying the unique effects of masked exposure to combat-related images (VBE) on the brain activity of U.S. combat veterans with PTSD. Study investigators will conduct a randomized controlled trial of VBE during fMRI scanning by manipulating awareness of exposure to combat-related stimuli, comparing the effects of VBE and (barely) visible exposure to these stimuli on the brain activity of 40 combat veterans with PTSD. Visible exposure to combat images is an active control condition that demonstrates the advantages of implicit exposure (VBE) in engaging extinction circuits and reducing fear responses. These advantages are not merely the consequences of exposure, but of how that exposure is delivered. The study thesis is that exposure is more effective, both in terms of circuit activity and fear responses, when delivered implicitly. Study investigators will manipulate the number of exposure sessions within each treatment group in order to identify the optimal number of sessions.
2. Directly relating the effects of VBE on neural activity to those on behavioral symptoms of PTSD. Subjective fear levels will be measured. In statistical analyses, changes in brain activity induced by VBE will be directly related to its ensuing effects on all of these measures, and the neural mechanisms that mediate the reduction of PTSD symptoms will thereby be inferred.

ELIGIBILITY:
Inclusion Criteria:

Patient Population

* Males and females ages 18-50
* Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) diagnosis of PTSD
* Traumatic event is a combat-based experience (e.g., being injured, watching a buddy be killed)
* Minimum score of 18 on the Combat Experience Scale (CES)
* Minimum score of 3 or more on Primary Care (PC)-PTSD-5
* Participants with other cooccurring psychiatric disorders (e.g., anxiety, ADHD) will be included to ensure a representative sample.

Healthy Population

• Males and Females, ages 18-50

Exclusion Criteria:

Patient Population

* Treatment for PTSD, substance abuse, or mental health concerns in the past 6 months
* 10 or more years since the combat trauma
* Acute intoxication
* Severe level of Substance Dependence (6 or more DSM-V symptoms)
* Prior diagnosis of Autistic Spectrum Disorders
* Current or past psychotic disorders or active psychotic symptoms
* Current Bipolar I Disorder
* Dementia
* Neurological or serious medical conditions (e.g., stroke, epilepsy/ seizure disorder, cancer, Lupus, HIV+);
* Traumatic brain injury

Healthy Population

* Ferromagnetic implants (e.g., pacemaker), metal braces, retainers, tattoos or permanent make up w/ metallic content, transdermal medicinal patches that cannot be removed
* Neurological or serious medical conditions (e.g., stroke, epilepsy/ seizure disorder, cancer, Lupus, HIV+);
* Lifetime Diagnosis of PTSD, Tourette's Syndrome, Bipolar Disorder, Substance Dependence, Eating Disorder, Autism Spectrum Disorder, a psychotic disorder, Acute Stress Disorder
* Lifetime history of traumatic event defined as a life-threatening event involving physical attack, guns, fire or explosion (i.e the kinds of traumatic events combat veterans are likely to experience)
* Traumatic Brain Injury
* Birth at less than 37 weeks gestational age
* Claustrophobia
* Anxiety Disorder, Mood Disorder, Substance Abuse Disorder, Adjustment Disorder in past 2 years
* Treatment for mental health concern in past 2 years
* Pregnant Females

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Mean Activation of Frontostriatal and Prefrontal Brain Regions to combat stimuli in PTSD | Day 2
  A hypothesis-driven, group-level analysis will test brain activity, measured as Blood Oxygen Level Dependent (BOLD) response, in 4 regions of interest while minimizing Type II error.

SECONDARY OUTCOMES:
Fear induced by exposure to combat stimuli in PTSD in veteran group as measured by fear scale | Day 2
  After each block of 10 combat stimuli trials, participants rate levels of fear on a 10-point, 1-10 visual analogue scale with these anchor point: "1 - No fear", "5 - Moderate but Tolerable Fear", and "10 - Very Intense Fear".
Fear induced by exposure to combat stimuli in PTSD in healthy participants as measured by fear scale | Day 2
  After each block of 10 combat stimuli trials, participants rate levels of fear on a 10-point, 1-10 visual analogue scale with these anchor point: "1 - No fear", "5 - Moderate but Tolerable Fear", and "10 - Very Intense Fear".
Fear induced by exposure to combat stimuli in PTSD in veteran group as measured by fear scale | Days 3-7
  After each block of 10 combat stimuli trials, participants rate levels of fear on a 10-point, 1-10 visual analogue scale with these anchor point: "1 - No fear", "5 - Moderate but Tolerable Fear", and "10 - Very Intense Fear".

CONTACTS AND LOCATIONS:
Overall Officials: Bradley M Peterson, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Brain Imaging Lab, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT06218381/ICF_000.pdf